CLINICAL TRIAL: NCT03576391
Title: Examining the Influence of Fatigue on Anticipatory Postural Adjustments of the Trunk Muscles and Movement-related Cortical Potentials in Healthy Subjects During a Rapid Arm Task Perturbation
Brief Title: The Influence of Fatigue on Trunk Motor Control and Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016/0951
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Muscle Fatigue; Mental Fatigue; Event-related Potentials
Keywords: Sensorimotor control; Feedforward; Physical Fatigue; Cognitive Fatigue; Event-related potentials
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Each participant will perform all 3 experimental conditions spread out over 2 test days. At test day 1 the control condition is performed. Test day 2 follows at least 5 days after the 1st one in order to make sure participants are physically and mentally recovered as the protocol at test day 1 might induce some physical or mental fatigue. On test day 2 the other 2 conditions are tested in a randomised order: either first the physical fatigue condition, followed by the cognitive fatigue condition or vice versa.
Who Masked: Outcomes Assessor
Masking Description: The researcher that will perform the EMG-analysis, i.e. onset determination of the various muscles that were measured, will be blinded for participant, condition and muscle during that process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control condition (Experimental): Control condition to assess whether the repetition of a RAM task without fatiguing task in between 2 repetitions affects trunk motor control and cortical movement preparation.
  Interventions: Behavioral: Control condition; Behavioral: Rapid Arm Movements
- Physical Fatigue condition (Experimental): Fatigue condition to assess whether a physical fatiguing task in between 2 RAM tasks affects trunk motor control and cortical movement preparation for the 2nd RAM.
  Interventions: Behavioral: Rapid Arm Movements; Behavioral: Physical fatigue condition
- Cognitive Fatigue condition (Experimental): Fatigue condition to assess whether a cognitive fatiguing task in between 2 RAM tasks affects trunk motor control and cortical movement preparation for the 2nd RAM.
  Interventions: Behavioral: Rapid Arm Movements; Behavioral: Cognitive fatigue condition

INTERVENTIONS:
Behavioral: Control condition — 45 minute rest while seated. Watching an animated movie, sleeping was not allowed.
  Arms: Control condition
Behavioral: Rapid Arm Movements — 2 blocks of 80 trials of RAM in either a forward (n = 40) or backward (n = 40) shoulder flexion direction and back to neutral as fast as possible, with maintaining extension in the elbow. Visual cues (arrows) indicated the movement direction.
Behavioral: Physical fatigue condition — 40 minutes rest while seated followed by static endurance tasks, i.e. modified Biering-Sörensen task and static abdominal curl task.
  Arms: Physical Fatigue condition
Behavioral: Cognitive fatigue condition — 45 minutes of a cognitively fatiguing condition consisting of a modified incongruent Stroop color-word task.
  Arms: Cognitive Fatigue condition

SUMMARY:
This study aims at examining the influence of both physically and cognitively induced fatigue on trunk motor control on the one hand and brain activity related to movement preparation on the other hand, in healthy adult subjects. Furthermore, a comparison between the effects of both types of fatigue will be made. For this purpose a motor control task will be performed and compared before and after 3 specific interventions: i.e. a control intervention, a physical task and a cognitive task. Muscle and brain activity will be measured during each motor control task.

It is hypothesised that motor control will not be altered after a control task, i.e. seated rest for 45 minutes. With regards to the physical fatigue condition, it is expected that trunk muscles will contract earlier after this task than before due to altered motor control. Cognitive fatigue is hypothesised to have similar underlying processes as physical fatigue, thus a similar earlier muscle contraction is also expected after cognitive fatigue.

Lastly, as both types of fatigue are expected to induce a similar effect on motor control no significant differences between cognitive and physical fatigue are hypothesised. However, it is possible that the magnitude of this effect differs between types of fatigue, i.e. that 1 of both types has a bigger effect on motor control than the other.

With regards to brain activity in preparation of a motor control task similar hypotheses are formulated: no effect of the control task on brain activity, earlier and possibly increased brain activity after both fatiguing tasks, and no differences between both types of fatigue besides a possible difference in magnitude of effect.

DETAILED DESCRIPTION:
September 2016 - January 2017. 16 healthy, adult male and female participants aged 18-45 were tested for 3 conditions on 2 separate days, i.e. a control condition on test day 1; a physical and cognitive fatiguing condition in randomised order on test day 2.

2 blocks of 80 rapid arm movements (RAM1 and RAM2) with the dominant arm were performed per condition, while electroencephalography (EEG) of the brain and surface electromyography (sEMG) of the Internal Oblique/Transversus Abdominis, External Oblique, Multifidus and Iliocostalis Lumborum pars Thoracis muscles were measured bilaterally. sEMG of the Anterior Deltoid muscle of the dominant arm was also measured. These RAM's were used to induce an internal perturbation to the postural balance of subjects and is an often used task in the study of trunk motor control. In between 2 blocks of the RAM the condition-specific interventions were given. The control condition consisted of RAM1 - 45 minute rest - RAM2; the physical fatigue condition consisted of RAM1 - 45 minute physical fatigue task - RAM2; the cognitive fatigue condition consisted of RAM1 - 45 minute cognitive fatigue task - RAM2.

The physical fatiguing task was a static endurance task for the paravertebral muscles, i.e. modified Biering-Sörensen task, followed by a static endurance task for the abdominal muscles, i.e. a static abdominal curl in 45° of trunk flexion while seated.

The cognitive fatiguing task was a modified incongruent Stroop color-word task for 45 minutes.

At the beginning of each test day several questionnaires were also administered to control for fatigue and physical activity, i.e. Checklist Individual Strength (CIS), Profile Of Mood States (POMS) and International Physical Activity Questionnaire (IPAQ).

January - February 2018. an additional 6 subjects were tested in order to increase the sample size of this study.

Statistical analysis will be performed to assess whether and to what extent both physical and cognitive fatigue might influence motor control as measured with EMG during RAM. Furthermore, the effect of both types of fatigue on cortical movement preparation will also be assessed based on the EEG measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects.

Exclusion Criteria:

* People with a history of pain or current pain
* severe pathologies
* traumata
* cardiorespiratory disorders
* neurological disorders
* vestibular disorders
* endocrinologic disorders
* psychiatric and cognitive disorders
* colour blindness
* sleeping disorders
* psychological disorders or major depressions
* major surgery to the spine or upper limbs
* clinically relevant malalignments and deformities
* malignancies
* substance abuse of alcohol or drugs
* consumption of analgesics without prescription 24 hours or with prescription two weeks before testing
* use of psychotropic medication
* extreme physical activities two days before testing
* professional athletes
* pregnant women or women < 1 year postnatally

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Trunk muscle EMG latency | 2 hours
  Latency of the activation onset of the trunk muscles on EMG compared to prime mover onset (Anterior Deltoid) in milliseconds.
Contingent Negative Variation | 2 hours
  A cortical EEG-potential that reflects movement preparation in the timeframe between a warning cue and a go cue in Volt.

SECONDARY OUTCOMES:
Visual Analogue Scale for Fatigue | 10 seconds for every measurement
  A self-reported rating by participants for experienced general fatigue, which was assessed at baseline, after every RAM and after the condition-specific interventions. Participants had to indicate on a horizontal axis of 10 cm how fatigued they were with at the left side of the axis (0) 'not fatigued at all' and on the right side of the axis (10) 'maximally fatigued/worst fatigue ever experienced'. The numeric score (0-10) was calculated by the researcher and was not visible for participants.
Rating of Perceived Exertion/Borg | 5 seconds for every measurement
  A self-reported rating by participants for assessing how fatiguing a specific task/intervention was. This was assessed after every RAM task and after the physical and cognitive fatigue tasks. This is a vertical scale ranging from 6 at the top (no exertion) to 20 at the bottom ('maximal exertion') of the scale. Participants saw both incremental numbers from 6-20 and descriptions at numbers 7 ('very very light'), 9 ('very light'), 11 ('reasonably light'), 13 ('quite heavy'), 15 ('heavy'), 17 ('very heavy'), 19 ('very very heavy'), 20 ('maximal exertion').
Checklist Individual Strength | 5 minutes at the beginning of each test day
  For this study the CIS-fatigue subscale scores were used in order to quantify the subjective amount of fatigue subjects were experiencing at the onset of each test session.
Profile Of Mood States-Short Form | 5 minutes at the beginning of each test day
  The POMS-Short Form questionnaire required subjects to rate 32 words on a five-point, Likert-type scale ranging from 0-4 (0 = not at all, 4 = extremely) in accordance with their state of mood at that moment. These thirty-two items were divided into four negative subscales and one positive subscale, the total score of a subject consists of the difference of the sum of the negative scales and the positive scale. This means the lower the total score, the higher the positive mood of the subject.
International Physical Activities Questionnaire | 15 minutes at the beginning of each test day
  The IPAQ was administered before each test session to question participants about the physical activities they performed during the last 7 days. This in order to control for week-to-week differences in physical exertion levels and in order to compare physical activity between subjects. Based on these scores 3 levels of physical activity could be determined with level 1 (low), 2 (moderate) and 3 (high) physical activity. These levels are calculated based on the amount of hours low, moderate and high exerting activities had been performed the last 7 days.
General questionnaire | 10 minutes at the beginning of test day 1
  Demographical and physical characteristics were questioned in a self-developed general questionnaire as well as educational/occupational levels, substance and medication use, general physical and mental health, and sleep quality and quantity of the week and night at the beginning of test day 1.
General questionnaire-Short | 10 minutes at the beginning of test day 2
  Only a short part of the General Questionnaire was repeated at the start of test day two. Demographic, physical and educational/occupational information would not alter between 2 test days, so these sections were unnecessary to question again at test day 2. Therefore a shorter version with only questions about substance and medication use since the previous test day, general physical and mental health, and sleep quality and quantity of the week and night before the test session was administered on test day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, PT, PhD, Principal Investigator — University Ghent
Locations (1):
- Vakgroep REVAKI (Ghent University - Ghent University Hospital), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared after completion of the study.